CLINICAL TRIAL: NCT03153410
Title: A Pilot Study of a GVAX Pancreas Vaccine (With Cyclophosphamide) in Combination With a PD-1 Blockade Antibody (Pembrolizumab) and a Macrophage Targeting Agent (CSF1R Inhibitor) for the Treatment of Patients With Borderline Resectable Adenocarcinoma of the Pancreas
Brief Title: Pilot Study With CY, Pembrolizumab, GVAX, and IMC-CS4 (LY3022855) in Patients With Borderline Resectable Adenocarcinoma of the Pancreas
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J1766; IRB00130267 (Other: JHMIRB)
Record Dates: First submitted 2017-05-11; First posted 2017-05-15 (Actual); Results first posted 2024-10-15 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas vaccine; immunotherapy; antibody; PD-1; IMC-CS4; Pembrolizumab; GVAX; Borderline Resectable; CY; Cyclophosphamide; Adenocarcinoma; Neoplasms
MeSH Terms: conditions — Pancreatic Neoplasms; Adenocarcinoma; Neoplasms | interventions — Cyclophosphamide; pembrolizumab; LY3022855

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4 (Experimental)
  Interventions: Drug: Cyclophosphamide; Drug: GVAX Pancreas Vaccine (GVAX); Drug: Pembrolizumab; Drug: IMC-CS4

INTERVENTIONS:
Drug: Cyclophosphamide — 200 mg/m^2, intravenous (IV) infusion
  Patients receive neoadjuvant immunotherapy consisting of cyclophosphamide and pembrolizumab on day 1, IMC-CS4 on days 1, 8, and 15, and GVAX on day 2 of Cycles 1 and 2 (3 weeks/cycle). Patients will then undergo pancreaticoduodenectomy 2-3 weeks later, followed by standard of care adjuvant chemotherapy at the discretion of the primary oncologist. Patients may then receive 4 cycles (3 weeks/cycle) of adjuvant immunotherapy (same regimen as Cycles 1 and 2). Disease free patients may receive an additional 12 booster cycles (3 weeks/cycle) of immunotherapy consisting of pembrolizumab on day 1 of all 12 booster cycles, as well as cyclophosphamide on day 1 and GVAX on day 2 of the 6th and 12th booster cycle.
  Other Names: CY; Cytoxan
Drug: GVAX Pancreas Vaccine (GVAX) — 5x10^8 cells, six intradermal (ID) injections
  Patients receive neoadjuvant immunotherapy consisting of cyclophosphamide and pembrolizumab on day 1, IMC-CS4 on days 1, 8, and 15, and GVAX on day 2 of Cycles 1 and 2 (3 weeks/cycle). Patients will then undergo pancreaticoduodenectomy 2-3 weeks later, followed by standard of care adjuvant chemotherapy at the discretion of the primary oncologist. Patients may then receive 4 cycles (3 weeks/cycle) of adjuvant immunotherapy (same regimen as Cycles 1 and 2). Disease free patients may receive an additional 12 booster cycles (3 weeks/cycle) of immunotherapy consisting of pembrolizumab on day 1 of all 12 booster cycles, as well as cyclophosphamide on day 1 and GVAX on day 2 of the 6th and 12th booster cycle.
  Other Names: PANC 10.05 pcDNA-1/GM-Neo and PANC 6.03 pcDNA-1/GM-Neo vaccine
Drug: Pembrolizumab — 200 mg, intravenous (IV) infusion
  Patients receive neoadjuvant immunotherapy consisting of cyclophosphamide and pembrolizumab on day 1, IMC-CS4 on days 1, 8, and 15, and GVAX on day 2 of Cycles 1 and 2 (3 weeks/cycle). Patients will then undergo pancreaticoduodenectomy 2-3 weeks later, followed by standard of care adjuvant chemotherapy at the discretion of the primary oncologist. Patients may then receive 4 cycles (3 weeks/cycle) of adjuvant immunotherapy (same regimen as Cycles 1 and 2). Disease free patients may receive an additional 12 booster cycles (3 weeks/cycle) of immunotherapy consisting of pembrolizumab on day 1 of all 12 booster cycles, as well as cyclophosphamide on day 1 and GVAX on day 2 of the 6th and 12th booster cycle.
  Other Names: MK-3475,; KEYTRUDA®
Drug: IMC-CS4 — 75 mg (dose level 1) or 100 mg (dose level 2), intravenous (IV) infusion
  Patients receive neoadjuvant immunotherapy consisting of cyclophosphamide and pembrolizumab on day 1, IMC-CS4 on days 1, 8, and 15, and GVAX on day 2 of Cycles 1 and 2 (3 weeks/cycle). Patients will then undergo pancreaticoduodenectomy 2-3 weeks later, followed by standard of care adjuvant chemotherapy at the discretion of the primary oncologist. Patients may then receive 4 cycles (3 weeks/cycle) of adjuvant immunotherapy (same regimen as Cycles 1 and 2). Disease free patients may receive an additional 12 booster cycles (3 weeks/cycle) of immunotherapy consisting of pembrolizumab on day 1 of all 12 booster cycles, as well as cyclophosphamide on day 1 and GVAX on day 2 of the 6th and 12th booster cycle.
  Other Names: LY3022855

SUMMARY:
The purpose of this study is to evaluate whether combining cyclophosphamide (CY), pembrolizumab, GVAX and IMC-CS4 is effective and safe in patients with borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
This was a single center, open label, pilot study to evaluate the safety and intratumoral immune response of neoadjuvant/adjuvant triplet immunotherapy: CY/GVAX, Pembrolizumab, and IMC-CS4 in patients with resectable or borderline resectable Pancreatic ductal adenocarcinoma.

Patients received the combination of CY/GVAX with pembrolizumab and IMC-CS4 following completion of standard neoadjuvant chemotherapy (with or without radiation). Immunotherapy agents were given prior to and after surgical resection.

Patients receive neoadjuvant immunotherapy consisting of cyclophosphamide and pembrolizumab on day 1, IMC-CS4 on days 1, 8, and 15, and GVAX on day 2 of Cycles 1 and 2 (3 weeks/cycle). Patients will then undergo pancreaticoduodenectomy 2-3 weeks later, followed by standard of care adjuvant chemotherapy at the discretion of the primary oncologist. Patients may then receive 4 cycles (3 weeks/cycle) of adjuvant immunotherapy (same regimen as Cycles 1 and 2). Disease free patients may receive an additional 12 booster cycles (3 weeks/cycle) of immunotherapy consisting of pembrolizumab on day 1 of all 12 booster cycles, as well as cyclophosphamide on day 1 and GVAX on day 2 of the 6th and 12th booster cycle.

ELIGIBILITY:
Inclusion Criteria:

* Have histologically or cytologically proven adenocarcinoma of the pancreas.
* Patient's acceptance to have a core biopsy.
* Presence of at least one measurable lesion.
* Must not have metastatic disease.
* Patients must have measurable disease, defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >20 mm with conventional techniques or as >10 mm with spiral CT scan. See Section 10.1.2 for the evaluation of measurable disease.
* Must have received last dose of stereotactic body radiotherapy no longer than 28 days prior to enrollment.
* Must have received last dose of chemotherapy at least 14 days or longer prior to entry into the study.
* Age >18 years.
* ECOG performance status 0-1.
* Patient's blood, kidney and liver function must within normal limits
* Must use an acceptable form of birth control while on study.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Currently is participating or has participated in a study using any investigational therapy within the past 28 days or is currently using an investigational device.
* Major surgery 28 days prior to study entry excluding minor procedures (dental work, skin biopsy, etc.), celiac plexus block, and biliary stent placement.
* Used any systemic steroids, immunosuppressant medications and anti-neoplastic treatment in the past 14 days.
* Prior treatment with immunotherapy agents (including, but not limited to: IL-2, interferon, anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, anti-OX-40, anti-CD40, or anti-CTLA-4 antibodies).
* Used any growth factors including, but not limited to, granulocyte-colony stimulating factor (G-CSF), GM-CSF, erythropoietin, within 14 days of study drug administration. Use of such agents while on study is also prohibited.
* Received any prophylactic vaccine within 14 days of first dose of study drug or received a live vaccine within 30 days of study treatment.
* Currently have or have history of certain study-specified heart, liver, kidney, lung, neurological, psychological, immune or other medical conditions.
* History of any autoimmune disease: inflammatory bowel disease, (including ulcerative colitis and Crohn's Disease), rheumatoid arthritis, systemic progressive sclerosis (scleroderma), systemic lupus erythematosus (SLE) autoimmune vasculitis (e.g., Wegener's Granulomatosis), CNS or motor neuropathy considered to be of autoimmune origin (e.g., Guillian-Barre Syndrome, Myasthenia Gravis, Multiple Sclerosis). Patients with thyroid disease will be allowed.
* Has history of (non-infectious) pneumonitis that required steroids, history or evidence of interstitial lung disease or active, non-infectious pneumonitis.
* Has a pulse oximetry < 92% on room air.
* Evidence of ascites on imaging.
* Requires the use of home oxygen.
* Have known history of infection with HIV, hepatitis B, or hepatitis C.
* Have been diagnosed with another cancer in the past 5 years (except for superficial bladder cancer, non-melanoma skin cancers, or a low grade prostate cancer not requiring therapy)
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Known or suspected hypersensitivity to GM-CSF, hetastarch, corn, dimethyl sulfoxide, fetal bovine serum, trypsin (porcine origin), yeast or any other component of GVAX pancreas vaccine.
* Pregnant or breastfeeding women.
* Positive pregnancy test during the study.
* Women sexually active with a fertile man and of childbearing potential unwilling or unable to use an acceptable method to avoid pregnancy for the entire study and for up to 120 days after the last dose of study drug.
* Unwilling or unable to follow the study schedule for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-09-27 (Actual); Primary Completion 2022-03-09 (Actual); Study Completion 2023-08-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana DeJesus, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 2 participants were excluded from analysis because they did not receive the study drug.
Groups:
- Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4: Cyclophosphamide: 200 mg/m^2, intravenous (IV) infusion GVAX: 5x10^8 cells, six intradermal (ID) injections Pembrolizumab: 200 mg, intravenous (IV) infusion IMC-CS4: 75 mg (dose level 1) or 100 mg (dose level 2), intravenous (IV) infusion
  Patients receive neoadjuvant immunotherapy consisting of cyclophosphamide and pembrolizumab on day 1, IMC-CS4 on days 1, 8, and 15, and GVAX on day 2 of Cycles 1 and 2 (3 weeks/cycle). Patients will then undergo pancreaticoduodenectomy 2-3 weeks later, followed by standard of care adjuvant chemotherapy at the discretion of the primary oncologist. Patients may then receive 4 cycles (3 weeks/cycle) of adjuvant immunotherapy (same regimen as Cycles 1 and 2). Disease free patients may receive an additional 12 booster cycles (3 weeks/cycle) of immunotherapy consisting of pembrolizumab on day 1 of all 12 booster cycles, as well as cyclophosphamide on day 1 and GVAX on day 2 of the 6th and 12th booster cycle.
Period: Overall Study
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Started (Started = enrolled and received at least one dose of study drug) | 9
Completed (Completed = Received 18 cycles of treatment) | 2
Not Completed | 7

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 7
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With a Treatment-related Immunologic Effect
Description: Treatment-related immunologic effect is defined as an 80% or greater increase in the number of CD8+ T cells (and at least 1.8 times the baseline median absolute deviation) in surgically resected tumor tissue in comparison to the baseline biopsy in subjects that received at least 1 dose of neoadjuvant combination immunotherapy and underwent a R0, R1, or R2 surgical resection.
Time Frame: 8 weeks
Population: 8/9 patients were included in the analysis because obtaining pre-treatment biopsy was not possible in one patient.
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 8
Participants | 6

2. Primary Outcome: Safety of the Combination of GVAX Pancreas Vaccine (With CY), Pembrolizumab, and a Macrophage Targeting Agent (CSF1R Inhibitor IMC-CS4) in Patients With Resectable or Borderline Resectable Pancreatic Cancer (BRPC) Prior to and Following Surgery
Description: Number of subjects that experienced a grade 3 or higher study drug related adverse event
Time Frame: 25 months
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 9
Participants | 2

3. Secondary Outcome: Overall Survival (OS)
Description: OS will be measured from date of first dose until death or end of follow-up (OS will be censored on the date the subject was last known to be alive for subjects without documentation of death at the time of analysis). Estimation based on the Kaplan-Meier curve.
Time Frame: 44 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 9
months | 20.4 [17.5 to NA] — NA Explanation: Upper bound confidence interval was not estimable due to insufficient number of events

4. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS is defined as time from fist dose of study drug to the date of progression or death. Subjects were censored at the date of last scan if alive at the time of analyses or if the subject's date of death was greater than 3 months after last scan. Estimation based on the Kaplan-Meier curve.
Time Frame: 37 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 9
months | 12.6 [7.3 to NA] — NA Explanation: Upper bound confidence interval was not estimable due to insufficient number of events

5. Secondary Outcome: Immune-related Objective Response Rate (irORR)
Description: Immune-related Objective Response Rate (irORR) is defined as the number of patients achieving a complete response (irCR) or partial response (irPR) based on immune related response criteria (irRC) following the study immunotherapy prior to surgical resection. Per irRC criteria, Complete Response (irCR) is the disappearance of all target lesions, Partial Response (irPR) is a decrease in tumor burden by 50% or greater.
Time Frame: Up to 10 weeks from baseline irRC read
Population: 7/9 patients were evaluable for assessment by irRC criteria
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 7
Participants | 0

6. Secondary Outcome: Surgical Resectability Rate
Description: Surgical resectability after neoadjuvant therapy as determined by the number of patients able to undergo surgical resection.
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 9
Participants | 9

7. Secondary Outcome: Pathologic Response Rate
Description: Pathologic response as determined by surgical margins status at the time of surgery and response to neoadjuvant treatment per surgical specimen assessment (participants with <10% residual viable tumor is reported).
Time Frame: 8 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
Number analyzed (Participants) | 9
Participants | 7

ADVERSE EVENTS:
Time Frame: Serious and Other (Not Including Serious) Adverse Events were evaluated for up to 25 months. All-cause mortality was evaluated for up to 44 months.
Arm/Group | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4
All-Cause Mortality (participants affected / at risk) | 7/9
Serious Adverse Events (participants affected / at risk) | 5/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4 (N=9)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Biliary anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Fever (General disorders) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cyclophosphamide, GVAX, Pembrolizumab and IMC-CS4 (N=9)
Alanine aminotransferase increased (Investigations) | 2 (3)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 4 (4)
Chills (General disorders) | 1 (1)
CPK increased (Investigations) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 4 (9)
Fatigue (General disorders) | 2 (3)
Fever (General disorders) | 4 (6)
Flu like symptoms (General disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1)
Nausea (General disorders) | 2 (2)
Papulopustular rash (Skin and subcutaneous tissue disorders) | 1 (2)
Periorbital edema (Skin and subcutaneous tissue disorders) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 4 (9)
Vaccine site, bruising (Skin and subcutaneous tissue disorders) | 1 (1)
Vaccine site, erythema (Skin and subcutaneous tissue disorders) | 9 (19)
Vaccine site, induration (Skin and subcutaneous tissue disorders) | 8 (9)
Vaccine site, pruritus (Skin and subcutaneous tissue disorders) | 8 (14)
Vaccine site, warmth (Skin and subcutaneous tissue disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 3 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Edema face (General disorders) | 1 (1)
Edema limbs (General disorders) | 1 (1)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Exocrine insufficiency (Gastrointestinal disorders) | 1 (1)
Headache (Nervous system disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Hypertension (Vascular disorders) | 2 (2)
COVID-19 Infection (Infections and infestations) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain in the rib cage (General disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Thrush (Infections and infestations) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1)
Weight loss (Investigations) | 4 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT03153410/Prot_SAP_000.pdf